CLINICAL TRIAL: NCT03412240
Title: Reverse RAMP Pacing to Terminate Ventricular Tachycardia ( REV-RAMP)
Acronym: REVRAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CD16/90568
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti tachycardia pacing (Experimental)
  Interventions: Procedure: Induced pacing of the heart

INTERVENTIONS:
Procedure: Induced pacing of the heart — Once the defibrillator leads have been inserted or, in the case of a box change, the old leads have been tested as per routine procedure, these pacing leads will be connected to an external pacing stimulator. The test involves electrically pacing your heart at different rates and we will be constantly monitoring you under close clinical supervision. During the test, your heart will be electrically stimulated to beat at a faster rate.

SUMMARY:
Cardiac pacing which involved stimulating the heart electrically with electrical wires that go into the heart is routine practice in the diagnosis and treatment of heart rhythm problems. Clinically this involved the fields of cardiac pacing and electrophysiology. Patients who are at risk of sudden death because of serious heart rhythms that are a result of malfunction of the electrical system of the pumping chambers of the heart (ventricles) are generally implanted with specialised pacemakers that can defibrillate (shock) the heart if a nasty life threatening rhythm should result. Shocks are painful and in order to try and treat these rhythms without shocks, anti tachycardia pacing is performed (this is routine part of the device), which aims to interrupt the rhythm by stimulating the heart electrically. This does not always work and can destabilise the rhythm leading to a shock. REVRAMP is a novel modification of anti tachycardia pacing which involved stimulating the heart through the defibrillator wires in a different way. It appears to work better and seems less likely to destabilise the heart rhythm, hence can reduce painful shocks.

DETAILED DESCRIPTION:
Cardiac pacing which involved stimulating the heart electrically with electrical wires that go into the heart is routine practice in the diagnosis and treatment of heart rhythm problems. Clinically this involved the fields of cardiac pacing and electrophysiology. Patients who are at risk of sudden death because of serious heart rhythms that are a result of malfunction of the electrical system of the pumping chambers of the heart (ventricles) are generally implanted with specialised pacemakers that can defibrillate (shock) the heart if a nasty life threatening rhythm should result. Shocks are painful and in order to try and treat these rhythms without shocks, anti tachycardia pacing is performed (this is routine part of the device), which aims to interrupt the rhythm by stimulating the heart electrically. This does not always work and can destabilise the rhythm leading to a shock. REVRAMP is a novel modification of anti tachycardia pacing which involved stimulating the heart through the defibrillator wires in a different way. It appears to work better and seems less likely to destabilise the heart rhythm, hence can reduce painful shocks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are due to have a new defibrillator (including cardiac resynchronisation defibrillator) implant or box change

Exclusion Criteria:

* Contraindications to defibrillator testing e.g. severe untreatable coronary disease Intracardiac thrombus Interruption of anticoagulation Participants undergoing box change, device upgrade or revision Inability or unwillingness to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Termination/cessation of ventricular tachycardia by rev ramp pacing protocol | 10 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom